CLINICAL TRIAL: NCT07126977
Title: The Effect of Video Game-Based Balance Exercises Added to Standard Rehabilitation on Clinical Symptoms and Pelvic Floor Muscle Functions in Children With Lower Urinary Tract Dysfunction
Brief Title: Video Game-Based Balance Training in Children With Lower Urinary Tract Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Tuğçe Oskay, Physiotherapist, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: -78097791-020-4281
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Lower Urinary Tract Dysfunction
Keywords: pelvic floor; lower urinary tract dysfunction; rehabilitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Virtual reality-assisted, video game-based balance exercises will be implemented in addition to the standard protocol for pelvic floor muscle rehabilitation. The exercise sessions will consist of a 5-minute warm-up period, 20 minutes of balance exercises, and a 5-minute cool-down period. All sessions will follow the same protocol, with the same game sequence and durations. Each game will be played for approximately 5 minutes. However, the number of repetitions for each game will vary depending on the participant's performance level.
  As a therapeutic tool, the Wii console, Wii Fit Plus game disc, and Wii Balance Board will be used. The selected exercise games will include Hula Hoop Plus, Penguin Slide, Soccer Heading, Table Tilt, Tightrope Walk, Ski Jump, and Step Up.
  Interventions: Behavioral: Urotherapy training; Other: Diaphragmatic Breathing Exercise; Other: Biofeedback-Assisted Pelvic Floor Muscle Exercises; Other: Video Game-Based Balance Exercise Training; Other: Functional Exercise Training
- Control group (Active Comparator): The pelvic floor rehabilitation program consists of urotherapy education, diaphragmatic breathing exercises, biofeedback-assisted pelvic floor muscle exercises, and functional exercises. All children and their parents participating in the study will receive urotherapy education prior to the PFMR interventions. The urotherapy session will last approximately 60 minutes. Diaphragmatic breathing exercises will be performed in 3 sets of 10 repetitions. No invasive procedures will be used during the biofeedback-assisted pelvic floor exercises. Exercises will begin lying down and progress as control improves. These exercises will be performed for a total of 20 minutes, consisting of 2-5 seconds of contraction followed by 5-10 seconds of relaxation. The program will also include exercises aimed at improving core stabilization, dynamic neuromuscular control, and pelvic mobility. Exercise selection, repetitions, and duration will be adjusted based on individual needs and progression.
  Interventions: Behavioral: Urotherapy training; Other: Diaphragmatic Breathing Exercise; Other: Biofeedback-Assisted Pelvic Floor Muscle Exercises; Other: Functional Exercise Training

INTERVENTIONS:
Behavioral: Urotherapy training — Standard urotherapy consists of five main components aimed at regulating lower urinary tract (LUT) function in children: education about LUT function and dysfunction, establishing healthy voiding habits and behavioral modifications, lifestyle recommendations such as balanced fluid intake and nutrition, monitoring of symptoms and voiding habits, and consistent caregiver support. In contrast, specific urotherapy focuses on treating particular LUT dysfunctions and includes interventions such as alarm therapy, pelvic floor training, biofeedback, neuromodulation, and clean intermittent catheterization. All children and their caregivers participating in our study will receive urotherapy training prior to the pelvic floor rehabilitation interventions. Each urotherapy session will last approximately 60 minutes.
Other: Diaphragmatic Breathing Exercise — The exercise will be performed under the supervision of a physiotherapist, twice a week for 8 weeks. After the correct position is established, participants will be instructed to slowly inhale through their nose and focus on feeling the breath move from top to bottom (cranial to caudal). They will be asked to hold their breath for a few seconds, then exhale slowly through pursed lips. Additionally, they will be reminded not to push only their abdomen upward while inhaling, but to feel the intra-abdominal pressure expanding evenly in all directions (360 degrees). This exercise will be performed in 3 sets of 10 repetitions.
Other: Biofeedback-Assisted Pelvic Floor Muscle Exercises — No invasive procedures will be performed. The physiotherapist will begin with external palpation of the perineal area to teach correct pelvic floor contractions without using accessory muscles. Once the patient masters this, animation-supported biofeedback exercises will start. If relaxation is insufficient, biofeedback will first target muscle relaxation.
  Using the NeuroTrac Myoplus Pro4 device, surface electrodes will be placed at 2 and 7 o'clock on the perineum, and the reference electrode on the right thigh. Exercises will start in a lying position and progress to sitting and standing as control improves. Each session will last about 20 min, with 2-5 s contractions followed by 5-10 s relaxations.
Other: Video Game-Based Balance Exercise Training — In our study, in addition to the standard protocol, virtual reality-supported video game-based balance exercises will be performed twice a week for 8 weeks. Each session will include a 5-minute warm-up, 20 minutes of balance exercises, and a 5-minute cool-down period. All sessions will follow the same protocol, with identical game order and duration. Each game will be played for approximately 5 minutes, and the number of repetitions for each game will vary depending on the participant's performance level.
  As a therapeutic tool, the Wii console, Wii Fit Plus game disc, and Wii Balance Board will be used. The selected exercise games will include Hula Hoop Plus, Penguin Slide, Soccer Heading, Table Tilt, Tightrope Walk, Ski Jump, and Step Up.
  Arms: Intervention group
Other: Functional Exercise Training — Our study will include exercises aimed at improving core stabilization, dynamic neuromuscular control, and pelvic mobility. Exercise selection will be tailored to individual needs, and the number of repetitions and duration will be adjusted based on the participant's progress. Preferred exercises will include movements such as bridge, dead bug, bilateral arm and leg lift, bear position, cat-camel, and pelvic clock.

SUMMARY:
This study aims to investigate the effects of video game-based balance exercises, in addition to standard treatment, in children aged 5-12 years with lower urinary tract dysfunction (LUTD). The single-center study will include 30 children who will be randomly assigned to an experimental group (video game-based balance exercises + standard treatment) or a control group (standard treatment only). Children in the experimental group will play selected balance games using the Wii console and Wii Balance Board twice a week for 8 weeks.

All participants will receive the standard program consisting of urotherapy, diaphragmatic breathing exercises, biofeedback-assisted pelvic floor muscle training, and functional exercises. Outcomes will be assessed using a Bladder Diary, uroflowmetry, ultrasonography for post-void residual urine, pelvic floor muscle activity with EMG, the Dysfunctional Voiding and Incontinence Symptoms Score Questionnaire(DVISS), quality of life with the Pediatric Incontinence Quality of Life Questionnaire (PinQ), balance tests, the McGill Core Endurance Test, and the Physical Activity Enjoyment Scale.

DETAILED DESCRIPTION:
The aim of this study is to incorporate balance exercises into the standard clinical protocol applied to children with lower urinary tract dysfunction (LUTD) and to implement them through video game-based exercises. This approach is expected to bring about positive changes in clinical symptoms and pelvic floor muscle functions. The video game-based balance exercise program will be conducted in addition to the child's routine treatment, twice a week for a total of 8 weeks at the same rehabilitation center. Each session will consist of a 5-minute warm-up, 20 minutes of balance exercises, and a 5-minute cool-down. All sessions will follow the same protocol, game sequence, and duration. Each game will be played for approximately 5 minutes, and the number of repetitions will vary depending on the participant's performance level.

As therapeutic tools, the Wii console, Wii Fit Plus game CD, and Wii Balance Board will be used. Selected exercise games will include Hula Hoop Plus, Penguin Slide, Soccer Heading, Table Tilt, Tightrope Walk, Ski Jump, and Step Up.

In the standard program, participants will receive urotherapy training, diaphragmatic breathing exercises, biofeedback-assisted pelvic floor muscle training, and functional exercise education.

This single-center study will include 30 children aged 5-12 years who have been diagnosed with LUTD. Participants will be randomly assigned to either the experimental group (n=15) or the control group (n=15). No interventional procedures (such as injections or vaccinations) will be performed during the study. Prior to participation, informed consent forms will be obtained from the parents of children who meet the inclusion criteria and voluntarily agree to take part in the study.

Demographic and clinical data of all participants will be collected using a Patient Follow-Up Form prepared by the researchers. To evaluate daily bladder function, parents will be asked to complete a 2-day Bladder Diary under supervision. Voiding function will be assessed by uroflowmetry, while post-void residual urine will be evaluated by a pediatric urologist using ultrasonography. Pelvic floor muscle activity will be measured by a physiotherapist using an EMG-supported device. The severity of LUTD will be determined using the Dysfunctional Voiding and Incontinence Symptoms Score Questionnaire(DVISS). Additionally, the child's quality of life will be evaluated with the Pediatric Urinary Incontinence Quality of Life Questionnaire (PinQ); balance will be assessed with the Pediatric Berg Balance Scale and the Single-Leg Balance Test on a Bosu Ball; core stability with the McGill Core Endurance Test; and enjoyment of the video game-based program with the Physical Activity Enjoyment Scale.

ELIGIBILITY:
Inclusion Criteria:

* Being between 5 and 12 years of age
* Having a diagnosis of "Lower Urinary Tract Dysfunction" made by a pediatric urologist according to the criteria defined by the ICCS
* Voluntary participation of both the parent and the child in the study

Exclusion Criteria:

* Having any neurologically based condition
* Presence of any condition in the parent or child that affects the ability to respond to the assessment tools (e.g., intellectual disability, developmental delay, cognitive problems)
* Having any physical impairment (orthopedic, structural, etc.) that prevents the use of Wii-Fit
* Presence of malformations or anatomical anomalies in the urinary tract system
* History of urological surgery
* Having constipation and/or fecal incontinence
* Previous participation in pelvic floor muscle rehabilitation
* Regular use of medication

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Patient Follow-up Form | At the beginning and at the end of the 8th week
  All participants' age (years), body weight (kg), and height (m) data will be recorded. For the measurement of body weight and height, devices manufactured by Seca will be used. Body mass index (BMI) will be calculated by dividing body weight by the square of height and will be expressed in kg/m².
  During face-to-face interviews, the pediatric urologist will obtain detailed information from the families and children regarding medication use, surgical history, cognitive and mental status, neurological or anatomical problems, and clinical symptoms.
  Clinical symptoms to be evaluated by the pediatric urologist will include urgency, frequency, straining, daytime incontinence, enuresis, urinary tract infection (UTI), hesitancy, pain during urination, intermittent voiding, feeling of incomplete bladder emptying, and voiding postponement behaviors.
  The results of all other assessment methods used in the study will also be recorded in this form.
Uroflowmetry | This test will be applied to all participants at the beginning of the study and at the end of the 8th week.
  Uroflowmetry is an essential test for children with lower urinary tract dysfunction (LUTD). It is easy to perform, non-invasive, and quick, providing important data such as voided volume, voiding time, maximum flow rate, curve pattern, and flow rate. In our study, uroflowmetry will be performed using a device manufactured by AYMED®.
  Before the clinical visit, parents will be informed that the child should consume an adequate amount of non-irritating fluids. They will also be instructed that excessive and rapid fluid intake should be avoided to ensure the child reaches the desired bladder fullness in a healthy manner.
  The test will be performed when the child feels the urge to void. If the child's feet do not reach the ground, a footstool will be placed under their feet to eliminate the possibility of pelvic floor muscle contraction due to lack of support.
Post-Void Residual (PVR) Urine Measurement | Measurements will be performed at baseline and at the end of the 8th week for all participating children.
  Post-void residual (PVR) urine is defined as the amount of urine remaining in the bladder after voiding. PVR is an important parameter for evaluating voiding dysfunction and is considered a risk factor for urinary tract infections (UTIs). The volume of PVR should ideally be measured within the first 5 minutes after voiding, and optimally within <1 minute.
  According to the standardization published by the International Children's Continence Society (ICCS), a PVR greater than 30 mL or more than 21% of bladder capacity is considered significant in children aged 4-6 years. In children aged 7-12 years, a PVR greater than 20 mL or more than 15% of bladder capacity is considered significant.
  In our study, PVR will be measured immediately after the uroflowmetry test by a pediatric urologist using a transabdominal ultrasound device (Telemed®) through the suprapubic region. This technique is preferred because it is non-invasive.
Bladder Diary | All children participating in our study will be asked to complete a detailed bladder diary with their parents for two consecutive days at baseline and again at the end of the 8th week.
  The bladder diary is one of the most valuable tools designed to assess lower urinary tract symptoms in daily clinical practice due to its simplicity and low cost. According to the standardization published by the International Children's Continence Society (ICCS), a minimum of 48-hour bladder diary should be completed when evaluating a child with lower urinary tract dysfunction (LUTD). The bladder diary includes data such as voiding frequency and volume, fluid intake, and drinking habits. In this diary, the child's voiding frequency, voided volume, fluid intake, and any episodes of daytime urinary incontinence will be recorded. Fluid intake and voided volume will be documented in milliliters (mL), and voiding duration will be recorded in seconds (s). Additionally, the child's sensation of urgency while voiding will be noted using categorical descriptors such as "none," "mild," "moderate," or "severe."
EMG - Pelvic Floor Muscle Activation Measurement | Measurements of all children participating in the study will be made at the beginning and at the end of the 8th week.
  Surface electromyography (sEMG) is a reliable and non-invasive method used to assess the function of the pelvic floor muscles by detecting motor unit action potentials and evaluating muscle contractions in real time. In our study, pelvic floor muscle activation of all participating children will be assessed by a physiotherapist using the NeuroTrac MyoPlus Pro4 device. All measurements will be conducted by the same physiotherapist.
  Prior to the measurement, children will be asked to completely empty their bladder. To prevent cross-talk, two surface electrodes will be placed on the perineal region at the 2 o'clock and 7 o'clock positions, and the reference electrode will be placed on the right thigh.
  Children will first be instructed on the correct contraction techniques, focusing on ventral and cranial pelvic floor muscle activation. Subsequently, each child will undergo a "Work-Rest Assessment" protocol lasting a total of 55 seconds using the same device.
Dysfunctional Voiding and Incontinence Symptoms Score (DVISS) Questionnaire | We will ask the parents of all children participating in our study to complete this questionnaire at baseline and at the end of the 8th week.
  This is one of the most commonly used assessment tools and has been adapted into Turkish. It was first developed and published in 2005 by Akbal and colleagues. This questionnaire is designed to identify lower urinary tract symptoms (LUTS) and assess the severity of these symptoms.
  The first 13 questions evaluate symptoms such as daytime urinary incontinence, enuresis, daily voiding frequency, and constipation, while the 14th question assesses the impact of these symptoms on the individual's quality of life. The total score of the questionnaire ranges from 0 to 35.
  According to research, a score of 8.5 or higher has been reported to detect lower urinary tract dysfunction with 90% sensitivity. A higher total score indicates more severe voiding dysfunction. In a study conducted by Tuygun et al., it was suggested that the DVSS may serve as a highly sensitive and non-invasive indicator that should be used before proceeding to invasive methods.
Pediatric Incontinence Questionnaire (PinQ) | All children participating in our study will be evaluated using this questionnaire at baseline and at the end of the 8th week.
  PIN-Q is the first continence-specific quality of life scale developed for the pediatric population. It was specifically designed for children and adolescents by Bower in 2006. The Turkish validity and reliability study of the questionnaire was conducted by Hanımeli R. in 2011.
  Originally, the PIN-Q consisted of 28 items across seven domains, including social relationships, self-esteem, family relationships, body image, independence, mental health, and the treatment process. In later studies, these domains were consolidated into two main groups: Internal (15 items) and External (5 items), reducing the total number of questions to 20.
  The questionnaire can be completed by children within 5 to 15 minutes. Each item is scored from 0 (never) to 4 (always), and the total score ranges from 0 to 80. Higher scores indicate lower quality of life. The physiotherapist will read the questions to the children, and parents will leave the room to prevent influence.
Pediatric Berg Balance Scale | This scale will be administered by the same physiotherapist to all children in our study at baseline and at the end of the 8th week.
  The Berg Balance Scale (BBS) was adapted for children in 2003 by Franjoine and colleagues and renamed the Pediatric Berg Balance Scale (PBBS). The Turkish validity and reliability study of the scale was conducted by Erden et al. in 2020. The PBBS consists of 14 items, each scored from 0 to 4, with a maximum total score of 56.
  A score between 0-20 indicates balance impairment, 21-40 reflects an acceptable balance level, and 41-56 suggests good balance ability. In the PBBS, the original BBS items have been reorganized in a functional sequence from easier to more difficult movements. The duration of static postures has been shortened and instructions simplified to suit children. During the assessment, a stopwatch will be used to measure time, a measuring tape to define distances, a chair with back and arm support for sit-to-stand tests, a step for stair-climbing assessment, and a small ball for the object-pickup test.
Single-Leg Balance Test on Bosu Ball | Participants will be evaluated by the same physiotherapist at baseline and at the end of the 8th week.
  The Bosu ball, with its unstable half-sphere shape, challenges postural control and is used as an effective tool for balance assessment, especially in children. Unstable surfaces activate the somatosensory system, adding extra demand on balance mechanisms and providing a valuable test condition for evaluating postural stability. Wallace et al. (2024) demonstrated that the Bosu ball significantly increases the center of gravity height compared to other devices, resulting in a wider and faster sway range.
  In our study, to assess dynamic balance with higher sensitivity, all participants will perform a single-leg standing test on the Bosu ball under both eyes-open and eyes-closed conditions, and the durations will be recorded in seconds.
McGill Core Endurance Test | Participants will be evaluated by the same physiotherapist at baseline and at the end of the 8th week.
  Although there is no definitive consensus on the evaluation of core stabilization, various assessment methods exist to measure components such as endurance, flexibility, motor control, strength, and function. Among the components of core stabilization, endurance tests are considered the most reliable measures, followed by flexibility, strength, motor control, and functional tests.
  In our study, we will assess static endurance, which is one of the core stabilization components. Following the protocols developed by McGill et al., four fundamental core endurance tests will be applied. The purpose of these tests is to evaluate individuals' ability to maintain specified static positions for as long as possible. The tests include the trunk flexor test, trunk extensor test, and side plank tests for both sides.
Exercise Enjoyment Scale | This scale will be completed by the children in the experimental group at the end of the 8th week.
  The Exercise Enjoyment Scale-8 is a unidimensional assessment tool consisting of 8 items designed to measure individuals' level of enjoyment during exercise. Using a bipolar scoring method ranging from 1 to 7, the scale evaluates participants' enjoyment, motivation, focus, and emotional responses throughout the exercise process.
  The scale was adapted into Turkish by Soylu et al. in 2023, with its strong psychometric properties confirmed. Its brevity and practical applicability make it suitable for use in large participant groups. This scale is an important tool for assessing the psychological effects of exercise and motivational processes.

CONTACTS AND LOCATIONS:
Overall Officials: Tuğçe Oskay, BSc, PT, Principal Investigator — Bahçeşehir Univ, Grad Sch of Health Sci, MSc Physiotherapy & Rehabilitation, Istanbul, Turkey; Tuğçe Tahmaz, PT, PhD, Study Director — Bahçeşehir Univ, Faculty of Health Sci, Physiotherapy & Rehabilitation Dept, Istanbul, Turkey
Locations (1):
- Tuğtepe Pediatric Urology and Surgery Clinic, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol
Supporting Information: Study Protocol
Time Frame: June 2025 - February 2026

REFERENCES:
- [Background] Kuwertz-Broking E, von Gontard A. Clinical management of nocturnal enuresis. Pediatr Nephrol. 2018 Jul;33(7):1145-1154. doi: 10.1007/s00467-017-3778-1. Epub 2017 Aug 21. PMID 28828529
- [Background] Bright E, Cotterill N, Drake M, Abrams P. Developing a validated urinary diary: phase 1. Neurourol Urodyn. 2012 Jun;31(5):625-33. doi: 10.1002/nau.21254. Epub 2012 Jan 24. PMID 22275270
- [Background] Van Batavia JP, Combs AJ. The Role of Non-invasive Testing in Evaluation and Diagnosis of Pediatric Lower Urinary Tract Dysfunction. Curr Urol Rep. 2018 Apr 6;19(5):34. doi: 10.1007/s11934-018-0784-1. PMID 29623450
- [Background] Zivkovic V, Lazovic M, Vlajkovic M, Slavkovic A, Dimitrijevic L, Stankovic I, Vacic N. Diaphragmatic breathing exercises and pelvic floor retraining in children with dysfunctional voiding. Eur J Phys Rehabil Med. 2012 Sep;48(3):413-21. Epub 2012 Jun 5. PMID 22669134
- [Background] Kilcik MH, Ozdemir F, Elmas AT. Effectiveness of game-based core exercise in children with non-neuropathic bladder dysfunction and comparison to biofeedback therapy. Low Urin Tract Symptoms. 2023 Jan;15(1):16-23. doi: 10.1111/luts.12467. Epub 2022 Nov 11. PMID 36366947
- [Background] Snijders CJ, Vleeming A, Stoeckart R. Transfer of lumbosacral load to iliac bones and legs Part 1: Biomechanics of self-bracing of the sacroiliac joints and its significance for treatment and exercise. Clin Biomech (Bristol). 1993 Nov;8(6):285-94. doi: 10.1016/0268-0033(93)90002-Y. PMID 23916048
- [Background] Duarte Nde A, Grecco LA, Franco RC, Zanon N, Oliveira CS. Correlation between Pediatric Balance Scale and Functional Test in Children with Cerebral Palsy. J Phys Ther Sci. 2014 Jun;26(6):849-53. doi: 10.1589/jpts.26.849. Epub 2014 Jun 30. PMID 25013281
- [Background] Kuru S, Calik BB, Kabul EG, Yigit M. The relationship between the functional status of the extremities and "core" stabilization in women with fibromyalgia. Reumatologia. 2024;62(6):412-420. doi: 10.5114/reum/194594. Epub 2024 Dec 24. PMID 39866308
- [Background] McGill SM, Childs A, Liebenson C. Endurance times for low back stabilization exercises: clinical targets for testing and training from a normal database. Arch Phys Med Rehabil. 1999 Aug;80(8):941-4. doi: 10.1016/s0003-9993(99)90087-4. PMID 10453772
- [Background] Franjoine MR, Gunther JS, Taylor MJ. Pediatric balance scale: a modified version of the berg balance scale for the school-age child with mild to moderate motor impairment. Pediatr Phys Ther. 2003 Summer;15(2):114-28. doi: 10.1097/01.PEP.0000068117.48023.18. PMID 17057441
- [Background] Erden A, Acar Arslan E, Dundar B, Topbas M, Cavlak U. Reliability and validity of Turkish version of pediatric balance scale. Acta Neurol Belg. 2021 Jun;121(3):669-675. doi: 10.1007/s13760-020-01302-9. Epub 2020 Feb 19. PMID 32077065
- [Background] Tuygun C, Sertcelik N, Bakirtas H, Cakici H, Cetin K, Imamoglu AM. Usefulness of a new dysfunctional voiding and incontinence scoring system in predicting treatment effect in children with voiding dysfunction. Urol Int. 2007;79(1):76-82. doi: 10.1159/000102919. PMID 17627174
- [Background] Akbal C, Genc Y, Burgu B, Ozden E, Tekgul S. Dysfunctional voiding and incontinence scoring system: quantitative evaluation of incontinence symptoms in pediatric population. J Urol. 2005 Mar;173(3):969-73. doi: 10.1097/01.ju.0000152183.91888.f6. PMID 15711352
- [Background] Chmielewska D, Stania M, Kucab-Klich K, Blaszczak E, Kwasna K, Smykla A, Hudziak D, Dolibog P. Electromyographic characteristics of pelvic floor muscles in women with stress urinary incontinence following sEMG-assisted biofeedback training and Pilates exercises. PLoS One. 2019 Dec 2;14(12):e0225647. doi: 10.1371/journal.pone.0225647. eCollection 2019. PMID 31790463
- [Background] Bauer SB, Nijman RJ, Drzewiecki BA, Sillen U, Hoebeke P; International Children's Continence Society Standardization Subcommittee. International Children's Continence Society standardization report on urodynamic studies of the lower urinary tract in children. Neurourol Urodyn. 2015 Sep;34(7):640-7. doi: 10.1002/nau.22783. Epub 2015 May 21. PMID 25998310
- [Background] Samijn B, Van Laecke E, Vande Walle J, Pascal A, Deschepper E, Renson C, Van den Broeck C. Uroflow measurement combined with electromyography testing of the pelvic floor in healthy children. Neurourol Urodyn. 2019 Jan;38(1):231-238. doi: 10.1002/nau.23836. Epub 2018 Oct 12. PMID 30311676
- [Background] Fuentes M, Magalhaes J, Barroso U Jr. Diagnosis and Management of Bladder Dysfunction in Neurologically Normal Children. Front Pediatr. 2019 Jul 25;7:298. doi: 10.3389/fped.2019.00298. eCollection 2019. PMID 31404146
- [Background] Pekbay Y, Ergin O, Topuz B, Sarikaya S, Acar ZZ, Irkilata HC, Dayanc M. The effects of pelvic floor muscle therapy on symptoms, voiding, and pelvic floor muscle activity parameters in children with overactive bladder. Neurourol Urodyn. 2019 Jun;38(5):1430-1442. doi: 10.1002/nau.24007. Epub 2019 Apr 20. PMID 31006136
- [Background] Toprak N, Sen S, Varhan B. The role of diaphragmatic breathing exercise on urinary incontinence treatment: A pilot study. J Bodyw Mov Ther. 2022 Jan;29:146-153. doi: 10.1016/j.jbmt.2021.10.002. Epub 2021 Oct 20. PMID 35248263
- [Background] Nieuwhof-Leppink AJ, Hussong J, Chase J, Larsson J, Renson C, Hoebeke P, Yang S, von Gontard A. Definitions, indications and practice of urotherapy in children and adolescents: - A standardization document of the International Children's Continence Society (ICCS). J Pediatr Urol. 2021 Apr;17(2):172-181. doi: 10.1016/j.jpurol.2020.11.006. Epub 2020 Nov 5. PMID 33478902
- [Background] Chang SJ, Van Laecke E, Bauer SB, von Gontard A, Bagli D, Bower WF, Renson C, Kawauchi A, Yang SS. Treatment of daytime urinary incontinence: A standardization document from the International Children's Continence Society. Neurourol Urodyn. 2017 Jan;36(1):43-50. doi: 10.1002/nau.22911. Epub 2015 Oct 16. PMID 26473630
- [Background] Pavione Rodrigues Pereira R, Nascimento Fagundes S, Surry Lebl A, Azevedo Soster L, Machado MG, Koch VH, Tanaka C. Children with nocturnal enuresis have posture and balance disorders. J Pediatr Urol. 2016 Aug;12(4):216.e1-6. doi: 10.1016/j.jpurol.2016.05.003. Epub 2016 May 20. PMID 27290613
- [Background] Austin PF, Bauer SB, Bower W, Chase J, Franco I, Hoebeke P, Rittig S, Walle JV, von Gontard A, Wright A, Yang SS, Neveus T. The standardization of terminology of lower urinary tract function in children and adolescents: Update report from the standardization committee of the International Children's Continence Society. Neurourol Urodyn. 2016 Apr;35(4):471-81. doi: 10.1002/nau.22751. Epub 2015 Mar 14. PMID 25772695
- See also: Quality of Life in Children with Urinary Incontinence and Their Families, and the Validity of the PinQ in Turkish Children — https://toad.halileksi.net/wp-content/uploads/2022/07/idrar-inkontinansli-cocuklarda-hastaliga-ozgu-yasam-kalitesi-olcegi-toad.pdf
- See also: Impact of Differing Instability Devices on Postural Sway Parameters — https://www.researchgate.net/publication/379593436_Impact_of_Differing_Instability_Devices_on_Postural_Sway_Parameters